CLINICAL TRIAL: NCT07246720
Title: Interpectoral-pectoserratus Plane Block vs. Serratus Posterior Superior Intercostal Plane Block for Postoperative Analgesia in Patients Undergoing Breast Cancer Surgery
Brief Title: IPP-PSP Block vs. SPSIPB in Breast Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Çağdaş Baytar, medical doctor, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025/16-9
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Acute Pain; Breast Cancer; Regional Anesthesia
Keywords: Interpectoral-Pectoserratus Plane Block; Serratus Posterior Superior Intercostal Plane Block; Breast Cancer Surgery; Opioid Consumption; Pain Management
MeSH Terms: conditions — Pain, Postoperative; Breast Neoplasms; Agnosia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group IPP-PSP (Active Comparator): Interpectoral-Pectoserratus Plane Block
  Interventions: Procedure: Interpectoral-Pectoserratus Plane Block
- Group SPSIPB (Active Comparator): Serratus Posterior Superior Intercostal Plane Block
  Interventions: Procedure: Serratus Posterior Superior Intercostal Plane Block

INTERVENTIONS:
Procedure: Interpectoral-Pectoserratus Plane Block — Ultrasound-guided injection between pectoralis major-minor and pectoralis minor-serratus anterior planes.
  Arms: Group IPP-PSP
Procedure: Serratus Posterior Superior Intercostal Plane Block — Ultrasound-guided injection between the serratus posterior superior muscle and the intercostal muscles.
  Arms: Group SPSIPB

SUMMARY:
This prospective, randomized clinical study aims to compare the analgesic efficacy of the interpectoral-pectoserratus plane block and the serratus posterior superior intercostal plane block for postoperative pain management in patients undergoing breast cancer surgery. Both techniques are ultrasound-guided regional anesthesia methods targeting different interfascial planes of the thoracic wall. The study will evaluate postoperative pain scores, opioid consumption, Quality of recovery and potential complications. The findings are expected to contribute to optimizing regional anesthesia strategies for enhanced recovery and improved analgesia following breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* ASA I-II-III risk groups
* Patients with informed consent
* Patients undergoing breast cancer surgery

Exclusion Criteria: • Ages <18 and >65

* ASA ≥ IV
* History of allergy to local anesthetics
* Known coagulation disorders
* Infection near the insertion site
* Chronic analgesic use
* Patients with diabetes mellitus and those receiving neoadjuvant chemotherapy (due to potential impairment of pain sensation)
* Body mass index >30
* Dementia or confusion
* Lack of cooperation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative opioid consumption | in the first 24 hours after completion of the surgical procedure
  Cumulative opioid consumption in the first 24 postoperative hours after the completion of the surgical procedure

SECONDARY OUTCOMES:
Postsurgical Quality of Recovery measured by the Quality of Recovery questionnaire | first day after surgery
  Postsurgical recovery by Quality of Recovery questionnaire (QoR-15) on first (D1) day after surgery.
  The minimum score on the Quality of Recovery questionnaire is 0 and the maximum score 150. Higher scores mean better quality of recovery.
Number of episodes of postoperative pain | In the first 24 hours after completion of the surgical procedure
  Number of episodes of postoperative pain (NRS score ≥ 4) at rest and at deep inspiration in the first 24 postoperative hours after the completion of the surgical procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguladk Bulent ecevit University, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No